CLINICAL TRIAL: NCT06367985
Title: CAPA-IVM Culture With Low Oxygen Tension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mỹ Đức Hospital (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03/24/DD-BVMD
Record Dates: First submitted 2024-03-26; First posted 2024-04-16 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: In Vitro Fertilization
Keywords: CAPA-IVM; Low Oxygen Tension; Oxygen; Culture; PCOS

STUDY DESIGN:
Intervention Model Description: Sibling oocytes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Air Oxygen Concentration CAPA-IVM culture (Experimental): Half of the COCs will be cultured in the CAPA step and IVM step at 37 degrees Celsius in air oxygen concentration (20%) and 6% carbon dioxide.
  Interventions: Other: Air Oxygen Concentration CAPA-IVM culture
- Low Oxygen Concentration CAPA-IVM culture (Active Comparator): Half of the COCs will be cultured in the CAPA step at a low oxygen concentration (5%) and IVM step at an air oxygen concentration (20%); all two steps combine 6% carbon dioxide at 37 degrees Celsius.
  Interventions: Other: Low Oxygen Concentration CAPA-IVM culture

INTERVENTIONS:
Other: Air Oxygen Concentration CAPA-IVM culture — * Group 1A: COC will be cultured in the CAPA step at an air oxygen concentration (20%) for 24 hours and 6% carbon dioxide at 37 degrees Celsius.
  * Group 1B: COCs will be cultured in the CAPA step at an air oxygen concentration (20%) for 24 hours and in the IVM step at an air oxygen concentration (20%) for 30 hours; all two steps combine 6% carbon dioxide at 37 degrees Celsius.
  Arms: Air Oxygen Concentration CAPA-IVM culture
Other: Low Oxygen Concentration CAPA-IVM culture — * Group 2A: COC will be cultured in the CAPA step at a low oxygen concentration (5%) for 24 hours and 6% carbon dioxide at 37 degrees Celsius.
  * Group 2B: COCs will be cultured in the CAPA step at a low oxygen concentration (5%) for 24 hours and the IVM step at an air oxygen concentration (20%) for 30 hours; all two steps combine 6% carbon dioxide at 37 degrees Celsius.
  Arms: Low Oxygen Concentration CAPA-IVM culture

SUMMARY:
Capacitation in-vitro maturation (CAPA-IVM) has recently been advanced in culturing oocytes from the germinal vesicle (GV) stage following mild or no controlled ovarian stimulation. Recent research suggested that O2 concentration may significantly regulate oocyte maturation and early embryo development through hypoxia-inducible factor (HIF). Nonetheless, it has been challenging to create the environmental culture conditions for addressing the optimal number of oocytes and the highest possibility of embryo development since consensus on the oxygen (O2) concentration index in the IVM culture environment has not been reached. Based on the outcomes of atmospheric O2 concentration (20%) and low O2 concentration (5%) during CAPA-IVM culture in mice, it has been hypothesized that a 5% O2 was the optimal culture condition for the pre-IVM step. A 20% O2 was more suitable for the IVM culture step. Therefore, this study is designed to enhance the CAPA-IVM culture system, improving treatment efficiency and providing various benefits for patients undergoing assisted reproductive technology.

DETAILED DESCRIPTION:
Capacitation in-vitro maturation (CAPA-IVM) has recently been advanced in culturing oocytes from the germinal vesicle (GV) stage. This approach is a modified version of conventional in vitro fertilization (IVF) and intracytoplasmic sperm injection (ICSI), following mild stimulation or no controlled ovarian stimulation occurred. Specifically, IVM can be indicated for patients diagnosed with polycystic ovary syndrome (PCOS), a higher number of secondary follicles (constituting nearly 15% of total patients), and treat a range of patients with the risks of ovarian hyperstimulation, venous thromboembolism or ovarian torsion. Additionally, CAPA-IVM helps shorten treatment time, is less expensive, and upgrades patient convenience without multiple follow-up examinations. The live birth rate after the first embryo transfer in the CAPA-IVM group was 35.2%, which was not statistically significantly different from the IVF group at 43.2% (risk difference -8.1%; 95% confidence interval from -16.6% to 0.5%). However, the number of high-quality embryos in each cycle and the cumulative clinical pregnancy rate in CAPA-IVM were still lower than in cIVF.

Moreover, further investigation should be considered due to the lack of high-quality evidence of concurrent reports. Therefore, improving the oocyte maturation conditions in CAPA-IVM to harvest the optimal number of oocytes and the highest possibility of embryo development is essential. Many studies conducted on both animal and human models have demonstrated that the effectiveness of CAPA-IVM depends on various factors. Among these, the environmental culture conditions such as oxygen (O2) concentration play a crucial role in producing healthy mature oocytes. O2 is a vital physical and chemical component of the fallopian tube, uterus and ovarian follicle, it is closely related to metabolic activity, oocyte maturation, and early embryo development. Recent research suggested that O2 concentration may significantly regulate oocyte maturation and early embryo development through hypoxia-inducible factor (HIF). A consensus on the O2 concentration index in the IVM culture environment has not been reached. Oocyte-embedded culture systems have been commonly used in two O2 concentrations, 5% and 20% worldwide. In the human body, cumulus-oocyte complexes (COCs) mature in conditions with low O2 concentrations ranging from 2% to 9%.

Conversely, COCs are exposed to an atmospheric O2 concentration of 20% during IVM manipulation and culture. Although the concentration of 5% mimics the most proper environment in the fallopian tube and uterus, the 20% O2 is widely applied in IVM techniques. The use of high concentrations facilitates a better progression of differentiation processes and increases the maturation rate of oocytes. However, some referential frames indicated that a 20% O2 may pose a risk of reactive oxidative stress (ROS), leading to an imbalance in the ratio of pro-oxidants to antioxidants, resulting in cellular damage. Furthermore, real-time respiration analysis of oocytes cultured at 5% O2 is similar to in vivo-developed oocytes but induced cellular activity and oxygen consumption at 20% O2. The impact of atmospheric O2 concentration (20%) and low O2 concentration (5%) during CAPA-IVM culture in mice shown in the study of Vrije Universiteit Brussel (VUB) - Belgium that the respiratory capability of COCs cultured at 5% O2 was relatively similar to COCs developing and maturing in vivo.

Nonetheless, COCs cultured at 20% O2 increased respiratory activity and oxygen consumption remarkably. The study observed that pre-IVM culture of COCs at 20% O2 caused developmental disruptions. Also, the result was unfavorable if mouse COCs were cultured at the IVM step with 5% O2. Based on these analyses, the researchers hypothesized that a 5% O2 was the optimal culture condition for the pre-IVM step, while a 20% O2 was more relevant to the IVM culture step. Combining these findings with results from VUB and characteristics of the differentiation process in CAPA-IVM oocytes, this study is divided into two main groups, including 5% pre-IVM and 20% IVM versus 20% pre-IVM and IVM) and demonstrates whether this hypothesis should be applied CAPA-IVM in human. The enhancement of the CAPA-IVM culture system leads to improved treatment efficiency of this technique and provides various benefits for patients undergoing assisted reproductive technology.

Study procedure:

Screening for eligibility

* This trial will be conducted at My Duc Hospital, Ho Chi Minh City, Viet Nam.
* Women who are potentially eligible will be provided information about the trial at the time of IVM treatment indication.
* Screening for eligibility will be performed on the day of the first visit when the IVM treatment is indicated.
* Patients will be provided information related to the study together with the informed consent documents. Signed informed consent forms will be obtained by the investigators from all women before the enrolment.

Oocytes will be divided into 2 groups:

Group 1 (includes 2 subgroups: 1A and 1B): Air Oxygen Concentration CAPA-IVM culture T = Total number of oocytes after OR and there are two subgroups.

The number of oocytes is divided below:

If T is an even number:

* Number of oocytes in Group 1A: One oocyte.
* Number of oocytes in Group 1B: T1B = (T-2)/2.

If T is an odd number:

* Number of oocytes in Group 1A: One oocyte.
* Number of oocytes in Group 1B: T1B = ([T-1]-2)/2. One oocyte remainder of the first patient will be assigned to group 1B, and the remainder of the next patient will be assigned to group 2B. Continuing to do so sequentially for the next remainder.

Group 2 (includes 2 subgroups: 2A and 2B): Low Oxygen Concentration CAPA- IVM culture T = Total number of oocytes after OR and there are two subgroups.

The number of oocytes is divided below:

If T is an even number:

* Number of oocytes in Group 2A: One oocyte.
* Number of oocytes in Group 2B: T2B = (T-2)/2.

If T is an odd number:

* Number of oocytes in Group 2A: One oocyte.
* Number of oocytes in Group 2B: T2B = ([T-1]-2)/2. One oocyte remainder of the first patient will be assigned to group 1B, and the remainder of the next patient will be assigned to group 2B. Continuing to do so sequentially for the next remainder.

Group 1A, 2A: Collecting after capacitation: oocyte and cumulus cell.

Group 1B, 2B: Collecting after capacitation: spent media, blank well. Collecting after maturation: spent media, cumulus cell, blank well.

ELIGIBILITY:
Inclusion Criteria:

* 18-42 years of age
* Diagnosed with polycystic ovary syndrome according to the Rotterdam criteria (2003)
* Indicating CAPA-IVM treatment
* Having at least 40 antral follicles in two ovaries by transvaginal ultrasound at the time of CAPA-IVM indication
* Agreeing to have frozen embryo transfer
* Agreeing to participate in the trial

Exclusion Criteria:

* Cycles with oocyte donation, preimplantation Genetic Testing (PGT)
* Couples with severe male factor (sperm concentration <5 million/ml, motility < 10%), surgical sperm retrieval
* Previous history of unexplained immature oocytes after IVF treatment
* Uterine abnormalities

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Maturation rate | Two day after oocyte retrieval
  The oocyte maturation rate was usually defined by MII oocyte number divided by total COCs number

SECONDARY OUTCOMES:
Total number of oocytes retrieval | On the day of oocyte retrieval
  Counting the number of oocytes retrieved
Number of patients with no oocyte retrieved | On the day of oocyte retrieval
  Counting the number of patients with no oocyte retrieved
Number of MII oocytes | Two day after oocyte retrieval
  The oocyte maturation was usually defined by MII oocyte number
Number of GV oocytes | Two day after oocyte retrieval
  Counting the number of GV oocytes
Number of patients with no matured oocyte | Two day after oocyte retrieval
  Counting the number of patients with no matured oocyte
Number of 2PN oocytes | 16-18 hours after ICSI
  Number of zygotes with 2 pronuclei after ICSI
Fertilization rate | 16-18 hours after ICSI
  Number of fertilized oocytes / number of oocytes inseminated
Abnormal fertilization rate | 16-18 hours after ICSI
  The percentage of zygotes with 1,3, or 4 pronuclei after ICSI / number of oocytes inseminated
Number of patients with no day-3 embryo | Five day after oocyte retrieval
  Counting the number of patients with no embryo
Number of day-3 embryos | Three days after intra-cytoplasmic sperm injection
  Counting the number of day-3 embryos at 64±2h after ICSI
Number of good quality Day-3 embryos | Three days after intra-cytoplasmic sperm injection
  Number of grade 1 and grade 2 day-3 embryos
Number of frozen day-3 embryos | Three days after ICSI
  Counting the numer of frozen day-3 embryos
Number of blastocyst (day 5 or day 6 embryo) | Five or six days after ICSI
  Counting the number of blastocyst at 114±2h/140±2h after ICSI
Number of patients with no blastocyst | Five or six days after ICSI
  Counting the number of patients with no blastocyst
Number of good quality blastocysts | Five days after intra-cytoplasmic sperm injection
  Number of grade 1 and grade 2 blastocysts
Number of frozen blastocysts | Three days after ICSI
  Counting the numer of frozen blastocysts
Number of embryos transferred | On the day of embryo transfer
  Total embryos transferred
Quality of embryos transferred (Grade 1, Grade 2, Grade 3) | On the day of embryo transfer
  The quality of transferred embryo is classified according to Alpha Scientists in Reproductive Medicine and ESHRE Special Interest Group of Embryology, 2011; D. Gardner, 1999; D. K. Gardner & Schoolcrati, 1999
Positive pregnancy test rate | 11 days after the day of blastocyst transfer and 13 days after the day of day-3 embryo transfer
  Positive pregnancy test defined as serum human chorionic gonadotropin level greater than 25 mIU/mL
Implantation rate | At 3 weeks after embryo transfer after the completion of the embryo transfer
  Implantation rate is explained as the number of gestational sacs per number of embryos transferred.
Clinical pregnancy rate | 5 weeks after embryo transfer
  Diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy at 6 weeks or more after the onset of last menstrual period. In addition to intra-uterine pregnancy, it includes a clinically documented ectopic pregnancy
Ectopic pregnancy rate | 3 weeks after embryo transfer
  A pregnancy outside the uterine cavity, diagnosed by ultrasound, surgical visualization or histopathology
Ongoing pregnancy rate | 10 weeks after embryo transfer
  Ongoing pregnancy is defined as pregnancy with a detectable heart rate at 12 weeks' gestation or beyond.
Miscarriage <12 weeks rate (Early miscarriage) | 2-10 weeks after embryo transfer
  Spontaneous loss of pregnancy up to 12 weeks of gestation is referred to as an early
Miscarriage <22 weeks rate (late miscarriage) | At >10 to 20 weeks after the transfer
  Spontaneous loss of pregnancy between 12 to 22 weeks is termed as late miscarriage
Live birth rate | At 22 weeks of gestation
  Live birth is defined as the complete expulsion or extraction from a woman of a product of fertilization, after 22 completed weeks of gestational age; which, after such separation, breathes or shows any other evidence of life, such as heartbeat, umbilical cord pulsation or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been cut or the placenta is attached. A birth weight of 500 grams or more can be used if gestational age is unknown. Twins counted as one live birth.
Multiple pregnancy rate | 4 weeks after embryo transfer
  Defined as the presence of more than one gestational sac at early pregnancy ultrasound (6-9 weeks gestation)
Multiple delivery rate | At 22 weeks' gestation
  Defined as the complete expulsion or extraction from a woman of more than one fetus, after 22 completed weeks of gestational age, irrespective of whether it is a live birth or stillbirth
Mode of delivery | At birth
  Vaginal delivery, C-section (elective, suspected fetal distress, non-progressive labor)
Gestational age at birth | At birth
  Calculated by gestational age of all live births
Birth weight | At the time of delivery
  in grams; of singletons and twins
Very low birth weight rate | At birth
  Birth weight less than 1.500 g
Low birth weight rate | At birth
  Birth weight less than 2.500 g
High birth weight rate | At birth
  Implies growth beyond an absolute birth weight, historically 4.000 g or 4.500 g, regardless of the gestational age
Very high birth weight rate | At birth
  Birth weight over than 4.500 g for women with diabetes, and a threshold of 5000 g for women without diabetes
Small for gestational age rate | At birth
  Large for gestational age was defined as a birth weight below the 10th percentile
Large for gestational age rate | At birth
  Large for gestational age was defined as a birth weight above the 90th percentile
Hypertension in pregnancy rate | At 20 weeks of gestation or beyond
  Comprising pregnancy-induced hypertension (PIH), pre-eclampsia (PET), eclampsia, and HELLP syndrome.
Gestational diabetes mellitus rate | At 24 to 28 weeks of gestation
  Diagnosed according to the latest version of ADA guidelines. a 75-g OGTT, with plasma glucose measurement when patient is fasting and at 1 and 2 h, at 24-28 weeks of gestation in women not previously diagnosed with diabetes.
  * Fasting: 92 mg/dL (5.1 mmol/L)
  * 1 h: 180 mg/dL (10.0 mmol/L)
  * 2 h: 153 mg/dL (8.5 mmol/L)
Still birth rate | After 20 completed weeks of gestational age
  defined as the death of a fetus prior to the complete expulsion or extraction from its mother after 20 completed weeks of gestational age. The death is determined by the fact that, after such separation, the fetus does not breathe or show any other evidence of life, such as heartbeat, umbilical cord pulsation, or definite movement of voluntary muscles. It includes deaths occurring during labor
Premature birth rate | On the day of delivery
  Defined as delivery at <24, <28, <32, <37 completed weeks. A birth that takes place after 22 weeks and before 37 completed weeks of gestational age.
Antepartum haemorrhage rate | At birth
  Defined as bleeding from or into the genital tract, occurring from 24 weeks of pregnancy and prior to the birth of the baby.
Major congenital abnormalities rate | At birth
  Structural, functional, and genetic anomalies, that occur during pregnancy, and identified antenatally, at birth, or later in life, and require surgical repair of a defect, or are visually evident, or are life-threatening, or cause death. Any congenital anomaly will be included as followed definition of congenital abnormalities in Surveillance of Congenital Anomalies by Division of Birth Defects and Developmental Disabilities, NCBDDD, Centers for Disease Control and Prevention (2020).
Neonatal mortality rate | between eight and 28 days after delivery
  Neonatal mortality defined as the death of a live-born baby within 28 days of birth. This can be divided into early neonatal mortality, if death occurs in the first seven days after birth, and late neonatal if death occurs between eight and 28 days after delivery
NICU admission rate | At birth
  Counting number of babies admited to neonatal intensive care unit
Reason for NICU admission | At birth
  Respiratory distress, Intraventricular Hemorrhage, Necrotizing enterocolitis, Sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vuong, MD, PhD, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Practice Committees of the American Society for Reproductive Medicine, the Society of Reproductive Biologists and Technologists, and the Society for Assisted Reproductive Technology. Electronic address: jgoldstein@asrm.org. In vitro maturation: a committee opinion. Fertil Steril. 2021 Feb;115(2):298-304. doi: 10.1016/j.fertnstert.2020.11.018. Epub 2020 Dec 24. PMID 33358333
- [Background] Paulson RJ, Fauser BCJM, Vuong LTN, Doody K. Can we modify assisted reproductive technology practice to broaden reproductive care access? Fertil Steril. 2016 May;105(5):1138-1143. doi: 10.1016/j.fertnstert.2016.03.013. Epub 2016 Apr 4. PMID 27054309
- [Background] Vuong LN, Ho VNA, Ho TM, Dang VQ, Phung TH, Giang NH, Le AH, Pham TD, Wang R, Smitz J, Gilchrist RB, Norman RJ, Mol BW. In-vitro maturation of oocytes versus conventional IVF in women with infertility and a high antral follicle count: a randomized non-inferiority controlled trial. Hum Reprod. 2020 Nov 1;35(11):2537-2547. doi: 10.1093/humrep/deaa240. PMID 32974672
- [Background] Gilchrist RB, Ho TM, De Vos M, Sanchez F, Romero S, Ledger WL, Anckaert E, Vuong LN, Smitz J. A fresh start for IVM: capacitating the oocyte for development using pre-IVM. Hum Reprod Update. 2024 Jan 3;30(1):3-25. doi: 10.1093/humupd/dmad023. PMID 37639630
- [Background] Zhao X, Liu X, Feng Y, Shi D, Lu F. Regulation of hypoxia-inducible factor 1alpha by optimal oxygen concentration enhances oocyte maturation and early embryonic development in buffalo. Theriogenology. 2023 Aug;206:50-59. doi: 10.1016/j.theriogenology.2023.05.006. Epub 2023 May 8. PMID 37187055
- [Background] Fischer B, Bavister BD. Oxygen tension in the oviduct and uterus of rhesus monkeys, hamsters and rabbits. J Reprod Fertil. 1993 Nov;99(2):673-9. doi: 10.1530/jrf.0.0990673. PMID 8107053
- [Background] Bahrami M, Cottee PA. Culture conditions for in vitro maturation of oocytes - A review. Reproduction and Breeding. 2022 Jun 1;2(2):31-6
- [Background] Increased susceptibility to oxidative stress as a proximate cost of reproduction - Alonso-Alvarez - 2004 - Ecology Letters - Wiley Online Library [Internet]. [cited 2023 Sep 19]. Available from: https://onlinelibrary.wiley.com/doi/10.1111/j.1461-0248.2004.00594.x
- [Background] Akin N, Ates G, von Mengden L, Herta AC, Meriggioli C, Billooye K, Stocker WA, Ghesquiere B, Harrison CA, Cools W, Klamt F, Massie A, Smitz J, Anckaert E. Effects of lactate, super-GDF9, and low oxygen tension during bi-phasic in vitro maturation on the bioenergetic profiles of mouse cumulus-oocyte complexdagger. Biol Reprod. 2023 Oct 13;109(4):432-449. doi: 10.1093/biolre/ioad085. PMID 37531262
- [Background] Herta AC, von Mengden L, Akin N, Billooye K, Coucke W, van Leersum J, Cava-Cami B, Saucedo-Cuevas L, Klamt F, Smitz J, Anckaert E. Characterization of carbohydrate metabolism in in vivo- and in vitro-grown and matured mouse antral folliclesdagger. Biol Reprod. 2022 Oct 11;107(4):998-1013. doi: 10.1093/biolre/ioac124. PMID 35717588
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS consensus workshop group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome (PCOS). Hum Reprod. 2004 Jan;19(1):41-7. doi: 10.1093/humrep/deh098. PMID 14688154